CLINICAL TRIAL: NCT03348735
Title: Safety, Efficacy and Patient Acceptability of Topical Treatment Versus Systemic Treatment: a Randomized, Multicentre, Comparative Pragmatic Trial in Adult Patients Suffering From Diverse Localized Neuropathic Pain (LNP) Syndromes
Brief Title: Localized Neuropathic Pain: Topical Treatment Versus Systemic Treatment
Acronym: PELICAN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low inclusion rate
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, Principle investigator, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R017007
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Capsaicin; Transdermal Patch; Pregabalin

STUDY DESIGN:
Intervention Model Description: A multicentre, randomized, open-label comparative trial evaluating topical treatment options (lidocaine 5% or capsaicine 8% patch) versus oral systemic treatment (pregabaline as standard of care) in adult patients suffering from localized neuropathic pain (LNP) syndromes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Stratified randomization by site and Neuropathic Pain Symptom Inventory (NPSI) will be applied, and coordinated centrally which randomizes eligible patients to one of three treatment arms, and assigns patient numbers. Medication will be dispensed by the hospital pharmacies of the individual participating multidisciplinary pain centres, after proper labelling.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lidocaine patch 5% (Experimental): Lidocaine 5% medicated plasters will be applied daily, during 12 consecutive hours.
  Interventions: Drug: Lidocaine patch 5%
- Capsaicin 8% patch (Experimental): Capsaicin 8% patches need to applied in a hospital setting during 1 hour. Re-application of these capsaicin patches will be performed upon re-occurrence of painful symptoms (mostly after 12 weeks - so not after a fixed time interval). Application of capsaicin patches will be carried out in a hospital setting (+/- 3 hours procedure).
  Interventions: Drug: Capsaicin 8% Patch
- Pregabaline (Active Comparator): Oral treatment with pregabalin (75mg capsules) will be used at optimized doses to best match clinical practice in Europe. In European clinical practice, up-titration of the dose is often carried out over a longer time-period. This study thus includes up-titration schedule for pregabalin over a period of 4 weeks. If patients develop side-effects during the intake/uptitration of pregabalin this treatment can be stopped and switched to gabapentin (300mg capsules). Gabapentin will always be the back-up treatment for failed systematic treatment with pregabalin. Dose of gabapentin will be uptitrated to maximum 1200mg per day.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Lidocaine patch 5% — Application of Lidocaine 5% patch for 12 hours.
  Arms: Lidocaine patch 5%
Drug: Capsaicin 8% Patch — Application of Capsaicin 8% patch for
  Arms: Capsaicin 8% patch
Drug: Pregabalin — Oral treatment with pregabalin (75mg capsules) will be used at optimized doses to best match clinical practice in Europe.
  Arms: Pregabaline

SUMMARY:
Evaluation of topical treatment with lidocaine 5% patch (daily administration) or capsaicin 8% patch (periodic administration - upon reoccurrence of pain symptoms) in adult patients suffering from localized neuropathic pain (LNP) across a wide variety of etiologies, with a duration between 1 and 24 months (subacute to chronic neuropathic pain (NP)).

DETAILED DESCRIPTION:
A multicentre, randomized, open-label comparative trial evaluating topical treatment options versus oral systemic treatment in adult patients suffering from localized neuropathic pain (LNP) syndromes. A wide variety of peripheral neuropathic pain syndromes will be included such as post-herpetic neuralgia (PHN), post-surgical NP/post-traumatic NP/scar pain, post-amputation NP, post-radiation therapy NP, complex regional pain syndrome (CRPS) type 1. In contrast to most (or even all) commercial clinical studies we will not limit the inclusion to one or two distinct neuropathic pain syndromes such as post-herpetic neuralgia (inclusion based on etiology of the neuropathic syndrome). In this pragmatic trial we will however include all patients suffering from a clinical neuropathic syndrome with distinct clinical features such as hyperalgesia/allodynia, presence of spontaneous positive sensory phenomena and lasting for more than 3 months without making any exclusion based on etiology. Initial pain intensity indicates the presence of either moderate or severe pain in these adult patients (NRS 4/10).

ELIGIBILITY:
Patients eligible for inclusion in this study must fulfil all of the following criteria:

* Subjects should be capable of giving their informed consent with sufficient knowledge of the Dutch, French or German language;
* Males and females, 18 years and older;
* Be assessed as suffering from moderate to severe neuropathic pain across the screening process with pain intensity (numeric rating scale - NRS) ≥ 4/10,
* At the time of screening pain symptoms have to be present for at least one (1) month, with a maximum of 24 months;
* Sensory disturbances present in the skin area of maximal pain;
* At the time of screening pain is clearly related to the presence of a localized neuropathic pain syndrome.
* Male or female patients of child producing potential* must agree to use contraception or take measures to avoid pregnancy during the study and until after the final treatment;
* Women can only be included after negative pregnancy test;

Exclusion Criteria:

* Age < 18;
* Pregnant and breastfeeding women;
* Infection in the painful skin region;
* Poorly healed or non-healed wound or scar in the painful skin region as well as presence of cutaneous abnormalities (non-intact skin barrier) within the painful skin region related to dermatological conditions;
* Known and/or strong suspicion of allergy to the study medication, known skin disorder (resulting in disruption of the normal skin barrier);
* Previous treatment with any of the three medications included in the study protocol for the same painful area within the last 12 months at the time of screening;
* Risk of heart failure and/or renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life questionnaire | 24 months
  To determine if topical treatment significantly improves health-related quality of life compared to systemic treatment in adult patients suffering from localized neuropathic pain across a wide variety of etiologies (LNP), with a duration between 1 and 24 months.

SECONDARY OUTCOMES:
Pain relief | from week 0 up to 26 weeks
  Reduction in pain intensity (PI-NRS), time to worsening of the pain (PI-NRS and NPSI) and use of rescue medication (MSQ III-R)
Health-related quality of life | from week 0 up to 26 weeks
  AUC for EQ-5D-5L measurements, global perceived effect (GPE), effect on mood (HADS), quality of sleep (NRS and ISI).
Drug tolerance | from week 0 up to 26 weeks
  Percentage of patients without systemic drug related side effects, percentage of patients who discontinue the study drug.
Functional status of the patient | from week 0 up to 26 weeks
  Impact of pain on functioning (Interference - BPI), participation in activities (Utrecht Work Engagement Scale), Work Productivity and Activity Impairment (WPAI).

CONTACTS AND LOCATIONS:
Overall Officials: Guy Hans, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (13):
- Belgium (13):
  - University hospital Antwerp, Edegem, Antwerp
  - AZ Monica (campus Antwerpen), Antwerp
  - AZ Klina, Brasschaat
  - AZ Sint Jan Brugge, Bruges
  - UVC Brugmann, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Ziekenhuis Oost-Limburg (ZOL, Genk
  - Universitair Ziekenhuis Gent (UZG), Ghent
  - UZ Brussel, Jette
  - Universitair Ziekenhuis Leuven (UZL), Leuven
  - Hopital Universitaire Sart Tilman de Liège (ULg) (CHU), Liège
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hans GH, Almeshal D, Vanlommel L, Roelant E, Verhaegen I, Smits E, Van Boxem K, Fontaine R, Investigators Team TP. Considerations on the Obstacles That Lead to Slow Recruitment in a Pain Management Clinical Trial: Experiences from the Belgian PELICAN (PrEgabalin Lidocaine Capsaicin Neuropathic Pain) Pragmatic Study. Pain Res Manag. 2023 Apr 14;2023:7708982. doi: 10.1155/2023/7708982. eCollection 2023. PMID 37089721